CLINICAL TRIAL: NCT03242304
Title: Changes in Plasma Cortisol, Brain-derived Neurotrophic Factor, and Nitrites in Patients With Acute Ischemic Stroke
Brief Title: Neuroactive Steroids in Acute Ischemic Stroke
Acronym: Cortisol
Status: Completed | Type: Observational
Sponsor: Hospital Militar Central, Argentina (Other)
Responsible Party: Principal Investigator, Sebastian Casas, Ph.D, M.D., Hospital Militar Central, Argentina
Other Study IDs: act No. 393 of Nov 11, 2015
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Ischemic Stroke; Cortisol; Hypersecretion
MeSH Terms: conditions — Ischemic Stroke | interventions — Behavior Rating Scale

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: A control group composed of subjects without physical or psychiatric disease.
  Interventions: Other: Behavioral tests
- Acute Ischemic Stroke group: An AIS group composed of subjects within the first 24 hours of the neurovascular event.
  Interventions: Other: Behavioral tests

INTERVENTIONS:
Other: Behavioral tests — We observed relationship between plasma levels of cortisol and neurological, cognitive, functional and emotional outcomes in patients with acute ischemic stroke.
  Other Names: Plasma cortisol levels quantification; Plasma nitrites levels quantification; Plasma Brain Derived Neurotrophic Factor quantification

SUMMARY:
Acute ischemic stroke (AIS) represents an economical challenge for health systems all over the globe. Despite increasing knowledge of the pathophysiology of AIS, there is no satisfactory treatment to revert the resulting brain damage. Changes of neuroactive steroids have been found in different neurological diseases. In this regard, the investigators have previously demonstrated that old patients with AIS show changes of plasma cortisol and estradiol concentrations, in that increased steroid levels are associated with a deterioration of neurological status and a worse cognitive decline. The present study assessed in patients with AIS if changes of behavior, brain-derived neurotrophic factor (BDNF) and nitrites (NO-2) (nitric oxide soluble metabolite) bear a relationship with the degree of hypercortisolism. To this purpose, the investigators recruited patients hospitalized at the Central Military Hospital emergency room within the first 24 hours of AIS. Subjects were divided into two groups, each one composed of 40 control subjects and 40 AIS patients, including men and women. The neurological condition was assessed using the NIHSS and the cognitive status with the Montreal Cognitive Assessment (MoCA test). The emotional status was evaluated using the Montgomery-Asberg Depression Rating Scale (MADRS), whereas the Modified Rankin Scale (MRS) was used to determine the functional condition. BDNF and NO-2 plasma levels were measured by ELISA and the Griess reaction method, respectively.

DETAILED DESCRIPTION:
Acute Ischemic Stroke (AIS) is one of the main causes of functional deterioration all over the world. Thus, 26% of patients older than 65 years still show limitations of daily activities 6 months after AIS, and 46% of these patients present cognitive deficiency of variable severity. AIS impose a burden on the way of living of patients and their families' in which depression emerges as a frequent neuropsychiatric disorder after the ischemic event. However, the occurrence of depression and other functional abnormalities on the first day following AIS is largely unknown. Neuroactive steroids have the capability to modulate in a positive or negative way the function of the nervous system. Changes in neuroactive steroid concentrations in plasma and nervous system have been described in degenerative diseases (Parkinson's disease, Alzheimer's disease, Huntington's disease, amyotrophic lateral sclerosis), autoimmune diseases (multiple sclerosis), epilepsy, and psychiatric disorders (depression and schizophrenia). In vulnerable regions such as the hippocampus and prefrontal cortex, high cortisol exposure damages the pyramidal neurons, decreases neurogenesis and impairs memory and learning. In a previous report, the investigators have demonstrated that old patients with AIS show changes in the plasma levels of cortisol and estradiol, which associate with low cognition, worse neurological status, and poor functional performance. The present report investigated changes of cortisol, brain-derived neurotrophic factor (BDNF) and nitrites (NO-2, nitric oxide soluble metabolites) after AIS. BDNF is a neurotrophin classically associated with learning and memory and negatively modulated by glucocorticoids, old age, and neurodegenerative diseases. In plasma, platelets are the major source of peripheral BDNF and levels of this neurotrophin are decreased in Alzheimer´s disease and depression. These disorders also show hypercortisolism and changes of cortisol dynamics suggesting that steroids, neurotrophins, and behavioral deficits may be functionally related. Regarding nitrites, cortisol treatment of human subjects significantly reduced plasma nitrate/nitrite concentrations. Therefore, considering that opposite changes occur in cortisol vs. BDNF and nitrites, the investigators aimed to determine in acute AIS patients (a) changes in plasma cortisol; (b) development of clinical, behavioral and functional deficits; (c) changes in plasma BDNF and nitrites, which may predict a neurotoxic effect of the excess cortisol in the ischemic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 90 years.
* Agreeing to participate in the study.
* Acute Ischemic Stroke of anterior vascular territory and/or posterior vascular territory whithin 24 hours of onset.
* Nine or more points in the Glasgow Coma Scale.
* Female patients in menopause.
* Patients without cognitive impairment before AIS according to family reference.
* Acceptance of the next of kin proxy in case the participant has sensory impairment.

Exclusion Criteria:

* Age <60 or > 90 years.
* Hemorrhagic Stroke.
* Transient ischemic attack (TIA).
* Acute Ischemic Stroke after 24 hours of onset.
* Hormonal replacement therapy.
* Immunosuppressive therapy in the last month before AIS (example corticosteroids).
* Acute infection (Example, pneumonia, urinary tract infection).
* Diagnosis of oncologic disease in the last month before AIS.
* Diagnosis of endocrinologic disease in the last month before AIS.
* Acute or long-term psychiatric illness.
* No agreement to participate in the study.
* Eight or less points in the Glasgow Coma Scale.
* Female patients with menstrual cycle or in the perimenopause.
* Patients with kidney or hepatic illness.
* Patients with cognitive impairment before AIS.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects were between 60 and 90 years old, and were recruited randomly and distributed in two experimental groups: 1) a control group composed of subjects without physical or psychiatric disease, 2) an AIS group composed of subjects within the first 24 hours of the neurovascular event. The individuals were distributed in such a way that each experimental group contained 10 men and 10 women. Table 1 show the inclusion and exclusion criteria used for the AIS group.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Neurological déficit | Into 24 hours of Acute Ischemic Stroke
  The neurological state during AIS was quantified by the National Institute of Health stroke scale at the time of hospitalization (NIHSS,available at http://www.ninds.nih.gov/doctors/NIH_Stroke_Scale.pdf

SECONDARY OUTCOMES:
Cognition | Into 24 hours of Acute Ischemic Stroke
  The cognitive test used was the Montreal Cognitive Assessment (MoCA test).
Emotional state | Into 24 hours of Acute Ischemic Stroke
  Patients with AIS were evaluated on the Montgomery-Asberg depression scale (MADRS)
Functional dependency of daily life activities | Into 24 hours of Acute Ischemic Stroke
  The functional state of the AIS patients was assessed by the modified Rankin scale at the time of entering the admission floor.
Cortisol | Into 24 hours of Acute Ischemic Stroke
  Plasma cortisol concentration was determined by chemiluminescent microparticle immunoassay (CMIA), using Team Architect i1000, Abbott Laboratories, Middletown, USA.
Quantification of nitrites concentration (NO-2) | Into 24 hours of Acute Ischemic Stroke
  Levels of NO-2, nitric oxide soluble metabolite (ON.) in water, were measured spectrophotometrically at 543 nm absorbance by the Griess reactio
BDNF quantification in plasma | Into 24 hours of Acute Ischemic Stroke
  Plasma BDNF concentration was measured by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian M Casas, Ph.D., MD., Principal Investigator — Hospital Militar Central Cir My ¨Dr. Cosme Argerich¨

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Casas S, Gonzalez Deniselle MC, Gargiulo-Monachelli GM, Perez AF, Tourreilles M, Mattiazzi M, Ojeda C, Lotero Polesel D, De Nicola AF. Neuroactive Steroids in Acute Ischemic Stroke: Association with Cognitive, Functional, and Neurological Outcomes. Horm Metab Res. 2017 Jan;49(1):16-22. doi: 10.1055/s-0042-119201. Epub 2016 Nov 3. PMID 27813048
- [Result] Yunes R, Casas S, Gaglio E, Cabrera R. Progesterone Exerts a Neuromodulatory Effect on Turning Behavior of Hemiparkinsonian Male Rats: Expression of 3 alpha -Hydroxysteroid Oxidoreductase and Allopregnanolone as Suggestive of GABAA Receptors Involvement. Parkinsons Dis. 2015;2015:431690. doi: 10.1155/2015/431690. Epub 2015 Mar 31. PMID 25918669
- [Result] Casas S, Giuliani F, Cremaschi F, Yunes R, Cabrera R. Neuromodulatory effect of progesterone on the dopaminergic, glutamatergic, and GABAergic activities in a male rat model of Parkinson's disease. Neurol Res. 2013 Sep;35(7):719-25. doi: 10.1179/1743132812Y.0000000142. Epub 2013 Mar 5. PMID 23561326
- [Result] Escudero C, Casas S, Giuliani F, Bazzocchini V, Garcia S, Yunes R, Cabrera R. Allopregnanolone prevents memory impairment: effect on mRNA expression and enzymatic activity of hippocampal 3-alpha hydroxysteroid oxide-reductase. Brain Res Bull. 2012 Feb 10;87(2-3):280-5. doi: 10.1016/j.brainresbull.2011.11.019. Epub 2011 Dec 6. PMID 22155686
- [Result] Ghersi MS, Casas SM, Escudero C, Carlini VP, Buteler F, Cabrera RJ, Schioth HB, de Barioglio SR. Ghrelin inhibited serotonin release from hippocampal slices. Peptides. 2011 Nov;32(11):2367-71. doi: 10.1016/j.peptides.2011.07.015. Epub 2011 Jul 27. PMID 21820473
- [Result] Casas S, Garcia S, Cabrera R, Nanfaro F, Escudero C, Yunes R. Progesterone prevents depression-like behavior in a model of Parkinson's disease induced by 6-hydroxydopamine in male rats. Pharmacol Biochem Behav. 2011 Oct;99(4):614-8. doi: 10.1016/j.pbb.2011.06.012. Epub 2011 Jun 15. PMID 21689676